CLINICAL TRIAL: NCT06148363
Title: Intervention Effect of High-Definition Transcranial Direct Current Stimulation (HD-tDCS) on Non-suicidal Self-injury (NSSI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Head, Dept of Neurology & Medical Psychology, Director, Cognitive Neuropsychology Lab, PRC, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHMU-tDCS-NSSI
Record Dates: First submitted 2023-11-19; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Transcranial Direct Current Stimulation; Non Suicidal Self Injury
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real stimulation (Active Comparator): The central electrode was placed over F3, with return electrodes at Fp1, Fz, F7 and C3. Fourteen 2-mA sessions (ramp-up and ramp-down periods of 15 and 15 seconds, respectively) were applied for 20 minutes per session, twice daily over 7 consecutive days.
  Interventions: Device: High-Definition transcranial Direct Current Stimulation (HD-tDCS)
- sham stimulation (Sham Comparator): In the sham condition, tDCS was delivered only during the ramp-up and ramp-down periods (15 and 15 s); no current was delivered during the 20-minute intervention. Participants will receive sham tDCS twice daily for two weeks.
  Interventions: Device: sham High-Definition transcranial Direct Current Stimulation (HD-tDCS)

INTERVENTIONS:
Device: High-Definition transcranial Direct Current Stimulation (HD-tDCS) — tDCS, or Transcranial Direct Current Stimulation, is a non-invasive brain stimulation technique that involves applying a small, constant direct current through electrodes placed on the scalp to modulate neuronal activity in specific brain regions.
  Arms: real stimulation
Device: sham High-Definition transcranial Direct Current Stimulation (HD-tDCS) — In the sham condition, tDCS was delivered only during the ramp-up and ramp-down periods (15s and 15s); no current was delivered during the 20-minute intervention.
  Arms: sham stimulation

SUMMARY:
To investigate the intervention effect of high-definition transcranial Direct Current Stimulation (HD-tDCS) on patients with Non-suicidal Self-injury (NSSI) and its underlying neural mechanism by magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Forty patients with Non-suicidal Self-injury (NSSI) diagnosed by DSM-5 were recruited from the Second Affiliated Hospital of Anhui Medical University. All participants underwent a structured interview and routine laboratory examination before and after receiving high-definition transcranial Direct Current Stimulation (HD-tDCS) treatment after meeting the inclusion criteria and obtaining informed consent. Each participant will complete the clinical evaluation, magnetic resonance imaging (MRI), and HD-tDCS treatment conducted by trained researchers at the Second Affiliated Hospital of Anhui Medical University. All the participants were randomized (1:1) to receive an "active HD-tDCS" or "sham HD-tDCS" treatment protocol. tDCS: the central electrode was placed over F3 with return electrodes placed at Fp1, Fz, F7 and C3. Fourteen 2-mA sessions (ramp-up and ramp-down periods of 15 and 15 seconds, respectively) were applied for 20 minutes per session, twice daily over 7 consecutive days. Sham HD-tDCS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 15 and 15 seconds.

Before and after the treatments, the patients received a battery measure of neuropsychological tests, and MRI scans in multimodalities. The neuropsychological assessment included the Ottawa Self-injury Inventory (OSI), the Adolescent Non-suicidal Self-injury Assessment Questionnaire (ANSAQ), the Hamilton Depression Rating Scale (HAMD), the Hamilton Anxiety Rating Scale (HAMA), and Patient Health Questionnaire-15 (PHQ-15), etc. Multimodal MRI includes 3D-T1, rs-fMRI, and DTI. The symptoms of the patients were followed up one and two months after the end of treatments.

ELIGIBILITY:
Inclusion Criteria:

The patients were diagnosed by 2 or more senior clinical psychiatrists, meeting DSM-V criteria, and having 1 or more non-suicidal self-injurious behaviors in the last 6 months.

12-18 years of age.

The medicine has not changed in the 4 weeks prior to or after this study, and if it has to be changed, the treatment medication is required to be at a subtherapeutic dosage level.

Exclusion Criteria:

The patient has suicidal ideation or has committed suicidal behavior

T1 or T2 weighted phase magnetic resonance images show focal brain lesions

patients had neurological disorders such as epilepsy, or serious physical illnesses

patients had a history of substance abuse and drug dependence in the last 6 months or use of anticonvulsant drugs in the last 3 months

patients had received radial cranial electrical stimulation or magnetic stimulation treatment in the last 3 months or received electroconvulsive therapy in the last 6 months

patients had previous significant head trauma or EEG abnormality in the last 1 month

body-mounted devices unsuitable for treatment, such as pacemakers, artificial valves, and other metal implants.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the number, frequency, and impulsivity of self-injurious behaviors | baseline and immediately after the intervention
  Adolescent Non-suicidal self-injury Assessment Questionnaire consisted of 2 dimensions and 12 items, with 5 options for each item, namely, "none, occasional, sometimes, often, and always", and was scored on a 5-point Likert scale from 0 to 4. The score for each item was summed up as the total score of the questionnaire, and the total mean score was divided by the number of items. The total mean score was divided by the number of items, and the higher the total mean score, the more serious the patients' non-suicidal Likert 5 self-injurious behaviors were.

SECONDARY OUTCOMES:
Change in Hamilton Depression Rating Scale (HAMD) Score | baseline and immediately after the intervention
  The HAMD is a clinician-administered depression assessment and consists of 17 items with a total score range from 0 to 54. A higher score indicates a worse outcome.
Change in Hamilton Anxiety Scale (HAMA) Score | baseline and immediately after the intervention
  The HAMA is a 14-item scale to measure the severity of anxiety symptoms, where each item is rated on a scale from 0 to 4. The HAMA total score ranges from 0 to 56, with lower scores indicating less anxiety symptoms.
Change in Patient Health Questionnaire-15 (PHQ-15) Score | baseline and immediately after the intervention
  The PHQ-15 is a 15-item scale to measure the severity of somatic symptoms, where each item is rated on a scale from 0 to 2. The PHQ-15 total score ranges from 0 to 30, with lower scores indicating less somatic symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China